CLINICAL TRIAL: NCT01165788
Title: Social Adaptation in Long Term Survivors of Blood and Marrow Transplantation
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BMT216; SU-07092010-6496 (Other: Stanford University)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Social Adaptation
Keywords: Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Social Adjustment

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- autologous BMT recipients: Lymphoma patients who received an autologous BMT as adults
  Interventions: Procedure: Semi structured personal interview

INTERVENTIONS:
Procedure: Semi structured personal interview — A trained research assistant will conduct in-person, in-depth semi-structured interviews at a location of the participants choosing. Participants will be asked to discuss their experiences with cancer, focusing especially on how their cancer affected their (1) work/education (2) relationships with their family (spouse, children, parents, siblings and other relatives) (3) their other social relationships

SUMMARY:
1. To explore specific aspects of social adaptation such as social connectedness, occupational outcomes and family relationships in lymphoma patients after autologous blood or marrow transplantation (BMT).
2. To investigate how social adaptation varies with time lapsed since BMT and with the life stage as determined by patient?s age. Understanding both the positive and negative aspects of cancer and cancer therapy leads to opportunities to promote adaptive strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Lymphoma patients treated with blood and marrow transplantation at Stanford University Medical Center
2. Age > 18 years at the time of transplant
3. English speaking
4. Willingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified from the comprehensive database of the Blood and Marrow Transplant Division of Stanford Hospitals & Clinics. We will target lymphoma patients who received an autologous BMT as adults (18 years or older). We estimate there are ~580 surviving who are between 2 and 22 years post-BMT.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Specific aspects of social adaptation, such as social connectedness, occupational outcomes and family relationships in lymphoma patients after autologous blood or marrow transplantation (BMT) | 1 year
Social adaptation variation with time lapsed since BMT and with the life stage as determined by patient's age | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cook, Principal Investigator — Stanford University; Kate Tierney, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States